CLINICAL TRIAL: NCT06745726
Title: Optimising Hypertension Management: Real-World Effectiveness of Zestril Personalised Dosing With the OptiZ Software as a Medical Device Companion App
Brief Title: OptiZ: Real World Evidence Study
Status: Not yet recruiting | Type: Observational
Sponsor: Closed Loop Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: CLM-HTN-006
Record Dates: First submitted 2024-12-13; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hypertension
Keywords: Hypertension; Zestril; lisinopril; mHealth; mobile app; self-monitoring; personalised medicine; blood pressure control; home blood pressure monitoring
MeSH Terms: conditions — Hypertension | interventions — Lisinopril

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single cohort: N/A, this is an observational study.
  Interventions: Drug: Zestril

INTERVENTIONS:
Drug: Zestril — N/A, this is an observational study.

SUMMARY:
Hypertension, or high blood pressure, is a major cause of preventable illness and premature death, affecting millions in the UK. Despite effective treatments, many patients struggle to achieve adequate blood pressure control. This study evaluates the effectiveness of the OptiZ. OptiZ is a mobile phone application ("app") intended to be installed on a mobile device as part of a treatment for hypertension for use by patients prescribed Zestril (lisinopril). The OptiZ app helps patients record blood pressure, dose-related side effects, and medication adherence, send reports to healthcare professionals for dose adjustments, set reminders to log their medication and blood pressure readings, and access information about high blood pressure and health tips.

This is a real-world observational study involving adults diagnosed with essential hypertension who are eligible for Zestril treatment. Recruitment will occur at selected GP practices across England over six months, with participants followed for 12 months. The study aims to enrol 113 participants. Using the OptiZ app, participants will record daily blood pressure readings, track medication adherence, record dose-related side effects, and access educational content on hypertension management. Healthcare professionals will use reports generated by the app to personalise Zestril dosing.

The main objective is to evaluate the OptiZ app's impact on reducing systolic blood pressure during the dose adjustment phase. Secondary objectives include adherence to Zestril, how often patients log blood pressure readings onto the OptiZ app and other patient-reported outcomes. Participants will also complete electronic questionnaires to provide feedback on their experience using the OptiZ app and their perceptions of hypertension treatment.

This study is funded by Closed Loop Medicine Ltd and Atnahs Pharma UK Ltd. The findings aim to improve hypertension care by using digital tools to enhance adherence, optimise dosing, and potentially reduce cardiovascular risks while guiding future digital solutions for chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years or older.
2. Participants must have a diagnosis of essential hypertension.
3. Participants must be eligible for Zestril prescription as part of their hypertension treatment plan, in line with the NICE stepwise approach, based on the clinical judgment of the responsible healthcare professional
4. Participants need to be willing to self-monitor, must be able to use a smartphone (iOS 16+ or Android 11+). A carer aged 18+ can use the app on their behalf if needed.
5. Participants must provide written informed consent to participate in the study, including agreeing to adhere to the study procedures.

Exclusion Criteria:

1. Participants with the following comorbidities: heart failure, a history of acute myocardial infarction, renal complications associated with diabetes mellitus, known clinically significant renal impairment (eGFR < 60 ml/min/1.73 m2). Participants with a strongly activated renin-angiotensin- aldosterone system (such as those with renovascular hypertension, salt and/or volume depletion, cardiac decompensation, or severe hypertension).
2. Participants with severe cognitive impairment or severe visual impairment/blindness that would prevent effective use of the smartphone app or self-monitoring using a blood pressure monitor (applies only if no carer is available).
3. Clinically significant abnormal blood results as judged by the responsible healthcare professional (including but not limited to, known abnormal serum potassium and/or blood urea nitrogen/serum creatinine renal).
4. Failure to satisfy the responsible healthcare professional of fitness to participate for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Uncomplicated primary hypertension cohort in England
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 12 months
  The change in systolic blood pressure from baseline to the end of the titration period.

SECONDARY OUTCOMES:
Mean change in diastolic blood pressure | 12 months
  Mean change in DBP from baseline to the end of titration period
Number and percentage of participants achieving target Home Blood Pressure at the end of their titration period | 12 months
  The number and percentage of participants achieving target HBP (home SBP [HSBP] less than 135 and home DBP [HDBP] less than 85 mmHg for adults aged under 80; below 145/85 mmHg for adults aged 80 and over) at the end of their titration period. with subsequent assessments at 4 months post successful titration and the end of the study (8-month follow-up).
Median time from baseline to first achieving Home Blood Pressure control | 12 months
  Median time from baseline to first achieving Home Blood Pressure control
Participants' daily adherence to Zestril | 12 months
  Participants' daily adherence to Zestril, assessed using the OptiZ App, with adherence success defined as adherence to prescribed medication on 80% or more days during the titration period.
Adherence to collecting data using the OptiZ App | 12 months
  Adherence to collecting data using the OptiZ App will be determined by the percentage of the titration period during which participants input data into the OptiZ App. Success will be defined as achieving 80% or more data input
Proportion of participants requiring re-entry into the titration phase at follow-up due to uncontrolled blood pressure | 12 months
  Proportion of participants requiring re-entry into the titration phase at follow-up due to uncontrolled blood pressure defined as home BP average of ≥135/85 mmHg for adults under 80 and ≥145/85 mmHg for those 80 and older.
Healthcare professionals' concordance to the OptiZ treatment report recommendations | 12 months
  Healthcare professionals' concordance to the OptiZ treatment report recommendations assessed using self-reported data via an e-questionnaire after each consultation visit with a participant
Participant's feedback using Brief Illness Perception Questionnaire | 8 months
  Participant's thoughts and emotions about treatment assessed using the Brief Illness Perception Questionnaire (B-IPQ) (consisting of 8 questions answered on a scale from 0 to 10 however each question is asked whereby a different a score of 0 or 10 is not consistently a better outcome; and a final question asking the participant to rank the 3 most important factors that they believe caused their illness) at baseline, end of titration period and 4-month follow up
Number and percentage of participants discontinuing Zestril due to unwanted side effects | 12 months
  Number and percentage of participants discontinuing Zestril due to unwanted side effects (or other clinically significant reasons as determined by the responsible healthcare professionals) assessed using data collected from medical notes and withdrawal forms
Number and type of spontaneously reported unwanted side effects | 12 months
  Number and type of spontaneously reported unwanted side effects, assessed using data reported during each consultation and from medical notes.
User experience and feedback on the OptiZ treatment | 8 months
  User experience and feedback on the OptiZ treatment assessed using the User Experience Questionnaire (UEQ) used to measure user experience with 6 scales (Attractiveness, Efficiency, Perspicuity, Dependability, Stimulation and Novelty) (where questions are answered on a scale from 1 to 7 but a score of 1 or 7 does not necessarily result in a better outcome). This questionnaires will be administered at the end of titration period and 4-month follow up.
User experience and feedback on the OptiZ treatment | 8 months
  User experience and feedback on the OptiZ treatment assessed using the UMUX-Lite questionnaire tailored to evaluate the specific components and features of the OptiZ App (consisting of 6 sections which all contain 2 questions where each question is answered using 'strongly agree', 'disagree', 'slightly agree', 'neither agree or disagree', 'slightly agree', 'agree', 'strongly agree' as well as a question for each section asking the participant why those scores were given). This questionnaires will be administered at the end of titration period and 4-month follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Oak Street Medical Practice, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No